CLINICAL TRIAL: NCT00584285
Title: Objective and Subjective Correlation Between Clinical Fluorescein Patterns and Theoretical Patterns Using the Medmont Corneal Topographer
Brief Title: Corneal Topographer Fluorescein Patterns
Status: Completed | Type: Observational
Sponsor: Christine Sindt (Other)
Responsible Party: Sponsor-Investigator, Christine Sindt, Asscociate Professor, University of Iowa
Organization: University of Iowa (Other)
Other Study IDs: 200709737
Record Dates: First submitted 2007-12-21; First posted 2008-01-02 (Estimated); Results first posted 2018-11-02 (Actual); Last update posted 2018-11-02 (Actual); Status verified 2018-03

CONDITIONS: Keratoconus
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Corneal Topographer Fluorescein Patterns: Use corneal topography to evaluate fluorescein pattern of rgp contact lens. Used corneal topography to develop theoretical fluorescein patters on a virtual eye. Theoretical lens developed by the topographer was ordered to compare to the actual fluorescein pattern on the actual eye.

SUMMARY:
The objective of this study is to determine if corneal topography can be used to predict the fluorescein pattern of keratoconus lenses on the eye. A corneal topography image will be taken and the computer selected lens will be placed on the eye. After placement of the lens color photographs will be taken of the eye's fluorescein pattern and compared to the computer predicted pattern.

DETAILED DESCRIPTION:
Subject population: keratoconus patients who have not undergone corneal surgery 100 subjects who come to UIHC for their contact lens care. We will approach them at their visit. We will not call potential participants from a database.

If topography is impossible to capture. Concommitant Corneal Disease Minors will be excluded

ELIGIBILITY:
Inclusion Criteria:

18 yrs of age or older with diagnosis of keratoconus and contact lens wearer

Exclusion Criteria:

Noncommittant corneal disease or surgery Inability to capture topography measurement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 18 yrs of age or older with diagnosis of keratoconus and contact lens wearer
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2007-09-15 (Actual); Primary Completion 2009-09-04 (Actual); Study Completion 2009-09-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine W. Sindt, OD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals and Clinics - Dept. of Ophthalmology, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Szczotka LB. Clinical evaluation of a topographically based contact lens fitting software. Optom Vis Sci. 1997 Jan;74(1):14-9. doi: 10.1097/00006324-199701000-00015. PMID 9148262
- [Background] Jani BR, Szczotka LB. Efficiency and accuracy of two computerized topography software systems for fitting rigid gas permeable contact lenses. CLAO J. 2000 Apr;26(2):91-6. PMID 10810939
- [Background] Rabinowitz YS, Garbus JJ, Garbus C, McDonnell PJ. Contact lens selection for keratoconus using a computer-assisted videophotokeratoscope. CLAO J. 1991 Apr;17(2):88-93. PMID 2049828
- [Background] Szczotka LB. Corneal topography and contact lenses. Ophthalmol Clin North Am. 2003 Sep;16(3):433-53. doi: 10.1016/s0896-1549(03)00054-3. PMID 14564765
- [Background] Bufidis T, Konstas AG, Mamtziou E. The role of computerized corneal topography in rigid gas permeable contact lens fitting. CLAO J. 1998 Oct;24(4):206-9. PMID 9800058

RESULTS

PARTICIPANT FLOW:
Groups:
- Corneal Topographer Flourscein Patterns: Use corneal topography to evaluate fluorescein pattern of rgp contact lens
  Comparison of fluorescein patterns: Compare trial contact lens fitting to fitting contact lenses based on corneal topography measurement
Period: Overall Study
Arm/Group | Corneal Topographer Flourscein Patterns
Started | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Corneal Topographer Flourscein Patterns: Use corneal topography to evaluate fluorescein patter of rgp contact lens
  Comparison of fluorescein patterns: Compare trial contact lens fitting to fitting contact lenses based on corneal topography measurement
Arm/Group | Corneal Topographer Flourscein Patterns
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 10
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With an Observable Difference Between Virtual Versus Actual Fluorescein Patterns
Description: Comparison of fluorescein patterns of rgp contact lens. Bearing and elevation fluorescein patterns will be compared between the actual (photo) and theoretical (computer generated) fluorescein patterns using standard clinical means.
Time Frame: Baseline first visit
Measure: Number; unit: participants
Groups:
- Corneal Topographer Flourscein Patterns: Use corneal topography to evaluate fluorescein pattern of rgp contact lens
  Comparison of fluorescein patterns: Compare conventional contact lens fitting to fitting contact lenses based on corneal topography measurement
Arm/Group | Corneal Topographer Flourscein Patterns
Number analyzed (Participants) | 18
participants | 0

ADVERSE EVENTS:
Groups:
- Corneal Topographer Flourscein Patterns: Use corneal topography to evaluate fluorescein pattern of rgp contact lens
  Comparison of fluorescein patterns: Compare trial lens contact lens fitting to fitting contact lenses based on corneal topography measurement
Arm/Group | Corneal Topographer Flourscein Patterns
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No